CLINICAL TRIAL: NCT01210976
Title: The Effects of Levosimendan on Haemodynamics in Patients Undergoing Elective Aortic Valve Replacement (AVR)Together With Coronary Artery Bypass Grafting
Brief Title: The Effects of Levosimendan on Haemodynamics in Patients Undergoing Elective Aortic Valve Replacement (AVR)Together With Coronary Artery Bypass Grafting (CABG) Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R08039M
Record Dates: First submitted 2010-09-24; First posted 2010-09-29 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Heart Valve Disease
Keywords: levosimendan; CABG; AVR
MeSH Terms: conditions — Heart Valve Diseases | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- levosimendan (Experimental)
  Interventions: Drug: levosimendan
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: levosimendan — 12 mcg/kg/10min bolus and 24 hour infusion at a rate of 0.2 mcg/kg/min
  Arms: levosimendan
Drug: placebo — nacl 0.9% coloured with thiamin in same volume and time than levosimendan
  Arms: placebo

SUMMARY:
Patients undergoing aortic valve replacement (AVR) surgery with coronary artery bypass grafting (CABG) are at risk of left ventricular dysfunction. The aim of the study is to describe the haemodynamic effects of levosimendan in comparison to placebo in patients undergoing elective aortic valve replacement (AVR) together with coronary artery bypass grafting (CABG) surgery. The study is randomized, double-blinded, placebo-controlled and will be carried out in Heart Center.

Twenty four patients will be randomized into two groups of 12. The treatment group will receive 24 hour infusion of levosimendan preoperatively where as the placebo group will receive an identical infusion of thiamine coloured glucose. The splanchnic perfusion will be measured by the means of vena hepatica cannulation. CircMon B202 (JR Medical Ltd, Tallinn, Estonia) is used for the measurement of whole-body impedance cardiography derived heart rate, cardiac index, left cardiac work index, systemic vascular resistance index (SVRI), and extracellular water (ECW). Surgical procedure, anaesthesia and cardio protection will be carried out as in standard care. Echo cardiography will be done pre- and postoperatively. Haemodynamics will be recorded hourly and mixed venous saturation every fourth hour for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* LVEF less than 50% of left ventricular hypertrophy indicated by wall thickness more than 12mm

Exclusion Criteria:

* allergy to levosimendan

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
blood pressure | up to 5 days

SECONDARY OUTCOMES:
echocardiography | baseline, 1st and 5th postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Heli Leppikangas, MD, Principal Investigator — Department of Anaesthesia, Tampere UH; Kati Järvelä, MD,PhD, Study Chair — Heart Center, Pirkanmaa Hospital District; Tero Sisto, MD, PhD, Study Chair — Heart Center, Pirkanmaa Hospital District; Pasi Maaranen, MD, Study Chair — Heart Center, Pirkanmaa Hospitla District; Pasi Lehto, MD,PhD, Study Chair — Heart Center, Pirkanmaa Hospital District; Marko Virtanen, MD,PhD, Study Chair — Heart Center, Pirkanmaa Hospital District; Sari Karlsson, MD, Study Chair — Department of Intensive Care, Tampere UH; Esko Ruokonen, MD,PhD, Study Chair — Department of Intensive Care, Kuopio UH; Leena Lindgren, MD,PhD, Study Director — Department of Anaesthesia, Tampere UH
Locations (1):
- Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Derived] Leppikangas H, Jarvela K, Sisto T, Maaranen P, Virtanen M, Lehto P, Karlsson S, Koobi T, Lindgren L. Preoperative levosimendan infusion in combined aortic valve and coronary bypass surgery. Br J Anaesth. 2011 Mar;106(3):298-304. doi: 10.1093/bja/aeq402. Epub 2011 Jan 21. PMID 21258075